CLINICAL TRIAL: NCT06516510
Title: A Randomised, Multi-centre, Intra-patient Imaging and Dosimetry Crossover Study of Lutetium (177Lu) rhPSMA-10.1 and Lutetium (177Lu) Vipivotide Tetraxetan (Pluvicto®) in Patients With Non-curative Metastatic Prostate Cancer
Brief Title: A Dosimetry Study of Lutetium (177Lu) rhPSMA-10.1 and Lutetium (177Lu) Vipivotide Tetraxetan (Pluvicto®) in Patients With Non-curative Metastatic Prostate Cancer
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Based on data from the Interim Analysis, the study will not adequately inform the clinical development programme for Lutetium (177Lu) rhPSMA-10.1 injection in the way that the study was intended. There are no concerns regarding participant safety.
Sponsor: Blue Earth Therapeutics Ltd (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: BET-PSMA-001
Record Dates: First submitted 2024-06-17; First posted 2024-07-24 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Lutetium; Lutetium-177; Pluvicto

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence A (Other): Patients in Sequence A will receive lutetium (177Lu) rhPSMA 10.1 followed by lutetium (177Lu) vipivotide tetraxetan
  Interventions: Drug: lutetium (177Lu) rhPSMA 10.1 and Pluvicto®
- Sequence B (Other): Patients in Sequence B will receive lutetium (177Lu) vipivotide tetraxetan followed by lutetium (177Lu) rhPSMA 10.1
  Interventions: Drug: lutetium (177Lu) rhPSMA 10.1 and Pluvicto®

INTERVENTIONS:
Drug: lutetium (177Lu) rhPSMA 10.1 and Pluvicto® — Radiopharmaceutical

SUMMARY:
A randomised, multi-centre, intra-patient imaging and dosimetry crossover study of lutetium (177Lu) rhPSMA 10.1 and lutetium (177Lu) vipivotide tetraxetan (Pluvicto®) in patients with non-curative metastatic prostate cancer

ELIGIBILITY:
Inclusion Criteria:

* Male patient aged ≥60 years old at Visit 1 (Screening).
* Patient has non-curative PSMA-positive prostate cancer that has spread outside of the prostate gland and is undergoing or being planned for radioligand therapy.
* At least 1 PSMA-positive lesion that can be outlined on PET or CT and ≥1 cm in the short axis measured on either modality, for the purpose of dosimetry.
* Adequate normal organ function as demonstrated by:

  * Absolute neutrophil count ≥1.5 × 109/L
  * Platelets ≥100 × 109/L
  * Haemoglobin ≥9 g/dL
  * Total bilirubin <2 × the institutional upper limit of normal (ULN). For patients with known Gilbert's Syndrome, ≤3 × ULN is permitted.
  * Alanine aminotransferase (ALT) or aspartate transaminase (AST) ≤3.0 × ULN or ≤5.0 × ULN for patients with liver metastases.
  * Estimated glomerular filtration rate (using Chronic Kidney Disease Epidemiology Collaboration Creatinine Equation [2009]) >50 mL/min.
* Willing to provide signed and dated written informed consent form (ICF) prior to any study specific procedures
* Male patients must agree not to father children or donate sperm during the study and for at least 14 weeks after the last study treatment.

Exclusion Criteria:

* Known hypersensitivity to lutetium (177Lu) rhPSMA 10.1 or lutetium (177Lu) vipivotide tetraxetan, or any of the constituents.
* Previous treatment with any radiopharmaceutical therapy in the 42 days or 5 half-lives prior to Visit 1 (Screening).
* Any significant metallic implants or objects, which may in the opinion of the investigator, affect image quality and/or dosimetry calculations.
* Severe claustrophobia, inability to lie flat or fit into the scanner, or any other inability to tolerate the SPECT/CT scan protocol
* Any change to prostate cancer medication or new prostate cancer therapy, prostate cancer surgical procedure within 42 days prior to screening or during the study.
* Any medical or psychiatric condition, including rapidly progressive prostate cancer, that in the investigator's judgment, makes the patient unsuitable for the study
* Participation in other studies involving other IMPs within 42 days or 5 half lives (whichever is longer) prior to Visit 1 (Screening) and/or during study participation

Min Age: 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
To compare the ratio of the kidney and the tumour absorbed doses of lutetium (177Lu) rhPSMA 10.1 and lutetium (177Lu) vipivotide tetraxetan. | 4-12 weeks

SECONDARY OUTCOMES:
To compare the absorbed dose of lutetium (177Lu) rhPSMA 10.1 and lutetium (177Lu) vipivotide tetraxetan to tumour lesions and additional organs of interest. | 4-12 weeks
To compare the tumour and normal organ effective half lives of lutetium (177Lu) rhPSMA 10.1 and lutetium (177Lu) vipivotide tetraxetan. | 4-12 weeks
To further evaluate the safety profile through frequency of treatment related adverse events of lutetium (177Lu) rhPSMA 10.1 injection | 4-12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Blue Earth Therapeutics, Study Director — Blue Earth Therapeutics
Locations (6):
- United States (2):
  - Biogenix Molecular LLC, Miami, Florida
  - Emory University Hospital, Atlanta, Georgia
- Radboud UMC, Nijmegen, Gelderland, Netherlands
- Spain (3):
  - Centro Integral Oncologico Clara Campal, Madrid, Madrid
  - Clinica Universidad de Navarra - Pamplona, Pamplona, Navarre
  - Clinica Universidad de Navarra, Madrid

IPD SHARING:
Plan to Share IPD: No